CLINICAL TRIAL: NCT06794879
Title: Survey of Parental Perception of Procedural Analgosedation in Pediatric Age.
Brief Title: Survey for Parental Perception of Procedural Analgosedation in Pediatric Age.
Acronym: ProSed-24
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ProSed-24
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Analgesia; Sensation, Hyperalgesic
Keywords: procedural analgosedation
MeSH Terms: conditions — Agnosia; Hyperalgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The conduction of this study may provide useful information about how much parents know and understand about procedural sedation, helping to identify any gaps. In addition, expectations and concerns about procedural sedation may be highlighted so that strategies aimed at improving communication by health care personnel can be developed. The results may guide the development of training programs for health care personnel so as to improve the management of procedural sedation and interaction with parents.

DETAILED DESCRIPTION:
The study involves the completion of a survey by Parents/Guardians, the remaining interventions will be performed following the normal care procedure outpatient regimen, according to normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children between the ages of 2 months and 14 years who are afferent to the withdrawal clinic

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children between the ages of 2 months and 14 years who are afferent to the withdrawal clinic of the U.O. Urgent Pediatrician, Emergency Department and Short and Intensive Observation of IRCCS - Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant'Orsola.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify the parent's degree of agreement/disagreement with pediatric procedural analgosedation practices and factors that may influence it | through study completion, an average of 1 year
  The parent's degree of agreement/disagreement with pediatric procedural analgosedation practices and the factors that may influence it will be analyzed by administering a survey

CONTACTS AND LOCATIONS:
Overall Officials: Laura Andreozzi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy, Italy